CLINICAL TRIAL: NCT05122195
Title: Effect of Graduated Elastic compRession Hosiery on vAricose Veins and Leg Edema in PrEgnant Women
Brief Title: Graduated Elastic compRession for vAricose Veins in PrEgnancy
Acronym: GRAPE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Belarusian State Medical University (Other)
Responsible Party: Principal Investigator, Vladimir Khryshchanovich, Professor, Belarusian State Medical University
Other Study IDs: 20140465
Record Dates: First submitted 2021-11-05; First posted 2021-11-16 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Varicose Veins; Pregnancy Related; Quality of Life
Keywords: VV's; GSV; SSV; QoL
MeSH Terms: conditions — Varicose Veins

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A, compression therapy group: Elastic compression therapy with a thigh length stockings of 23-32 mmHg, at least 8 hours a day.
  Interventions: Other: Compression therapy
- Group B, control group: No compression therapy prescribed in the follow-up period.

INTERVENTIONS:
Other: Compression therapy — Graduated elastic compression promote venous flow which is impaired by hormonal changes in the venous system during the gestational period and minimize the blocking effect of the gravid uterus.
  Groups: Group A, compression therapy group

SUMMARY:
This study will be evaluate the clinical efficacy of using graduated compression hosiery for venospecific symptoms, leg edema, and quality of life (QoL) in pregnant women with varicose veins (VV's).

DETAILED DESCRIPTION:
Each pregnant woman randomly receive an envelope. Those who received numbers 01 to 40 constitute the intervention group, and those with numbers 41 to 80 are in the control group.The intervention group will use a thigh length stockings with a compression of 23-32 mmHg, at least 8 hours a day. Verbal and written instructions on the proper use of the stockings will provide. During follow-up period, monitoring the regular use of compression stockings are performed every week. The physical characteristics of the patients, including the age, height, weight, and gestational week, are obtained and recorded. The clinical evaluation are performed using clinical-etiological and anatomical-pathophysiological assessment based on the CEAP classification.

Clinical examinations, QoL assessment and duplex-ultrasound will perform two qualified physicians in the 160 lower limbs of the 80 pregnant women with VV's at three landmark periods: between the 12th and 15th (initial examination), 20th and 28th (intermediate examination), and between the 28th and 36rd (final examination) week of gestation. The study protocol includes examination of the deep and superficial venous system with recording the reflux time and great and small saphenous veins (GSV/SSV) diameters in seven preestablished points, 5 points in the GSV and 2 points in the SSV. A reflux time in the superficial veins above 0.5 s is considered pathological reflux.

The ankle and lower leg circumference are measured using a measuring tape. Measurements are carried out at the lateral and medial ankle and the middle of the lower leg. All measurements are carried out at the same time of the respective days in the late afternoon or early evening; before the measurements the patients underwent a 45-min temperature and cardiovascular equilibrium period in a sitting position.

The QoL and subjective symptoms: tired, heavy legs, sensation of tension, tingling, and pain are assessed at each visit before the volume measurements and ultrasonographic evaluation. The subjective symptoms are evaluated by use of a semiquantitative scale from 0 to 3: 0 = no symptoms; 1 = mild; 2 = moderate; and 3 = severe. The QoL is investigated at each visit by a Chronic Venous Insufficiency Questionnaire (CIVIQ).

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women who are between the 12th and 15th weeks of gestation.
2. Primary symptomatic varicose veins, Clinical Etiological Anatomical Pathophysiological (CEAP) classification, clinical class C1-C3.
3. Ability to comprehend and sign an informed consent document.

Exclusion Criteria:

1. Deep venous thrombosis, thrombophilia associated with a high risk of deep venous thrombosis or postthrombotic syndrome.
2. Postoperative varicose vein disease recurrence.
3. History of pulmonary embolism.
4. Current compression therapy (within 7 days of enrollment).
5. CEAP clinical class C4-C6.
6. Arterial occlusive disease and lymphatic pathology of lower limbs.
7. Edema of limbs other than of venous origin.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women (between the 12th and 15th weeks of gestation) with primary varicose vein disease and C1-C3 are included in the prospective consecutive case study if they satisfied the selection criteria.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
Responders to Treatment, Assessed by Duplex Ultrasound | 8 weeks
  Responders; Number of Participants with eliminated superficial pathological reflux between the 20th and 28th weeks of gestation
Responders to Treatment, Assessed by Duplex Ultrasound | 16 weeks
  Responders; Number of Participants with eliminated superficial pathological reflux between the 28th and 36th weeks of gestation
Number of Participants with reduction of the GSV and SSV diameters, Assessed by Duplex Ultrasound | 8 weeks
  Responders; reduction of the GSV and SSV diameters between the 20th and 28th weeks of gestation
Number of Participants with reduction of the GSV and SSV diameters, Assessed by Duplex Ultrasound | 16 weeks
  Responders; Number of Participants with reduction of the GSV and SSV diameters between the 28th and 36th weeks of gestation
Responders to Treatment, Assessed by a measuring tape | 8 weeks
  Responders; Number of Participants with reduction of the ankle and lower leg circumference between the 20th and 28th weeks of gestation
Responders to Treatment, Assessed by a measuring tape | 16 weeks
  Responders; Number of Participants with reduction of the ankle and lower leg circumference between the 28th and 36th weeks of gestation
Number of Participants with pain from absent (score 0) to severe (score 3) | 8 weeks
  None (0), Occasional (1), Daily, intefering with, but not preventing daily activities (2), Daily, limiting most daily activities (3)
Number of Participants with pain from absent (score 0) to severe (score 3) | 16 weeks
  None (0), Occasional (1), Daily, intefering with, but not preventing daily activities (2), Daily, limiting most daily activities (3)
Number of Participants with heavy legs from absent (score 0) to severe (score 3) | 8 weeks
  None (0), Occasional (1), Daily, intefering with, but not preventing daily activities (2), Daily, limiting most daily activities (3)
Number of Participants with heavy legs from absent (score 0) to severe (score 3) | 16 weeks
  None (0), Occasional (1), Daily, intefering with, but not preventing daily activities (2), Daily, limiting most daily activities (3)
Number of Participants with tired legs from absent (score 0) to severe (score 3) | 8 weeks
  None (0), Occasional (1), Daily, intefering with, but not preventing daily activities (2), Daily, limiting most daily activities (3)
Number of Participants with tired legs from absent (score 0) to severe (score 3) | 16 weeks
  None (0), Occasional (1), Daily, intefering with, but not preventing daily activities (2), Daily, limiting most daily activities (3)
Number of Participants with sensation of tension from absent (score 0) to severe (score 3) | 8 weeks
  None (0), Occasional (1), Daily, intefering with, but not preventing daily activities (2), Daily, limiting most daily activities (3)
Number of Participants with sensation of tension from absent (score 0) to severe (score 3) | 16 weeks
  None (0), Occasional (1), Daily, intefering with, but not preventing daily activities (2), Daily, limiting most daily activities (3)
Number of Participants with tingling from absent (score 0) to severe (score 3) | 8 weeks
  None (0), Occasional (1), Daily, intefering with, but not preventing daily activities (2), Daily, limiting most daily activities (3)
Number of Participants with tingling from absent (score 0) to severe (score 3) | 16 weeks
  None (0), Occasional (1), Daily, intefering with, but not preventing daily activities (2), Daily, limiting most daily activities (3)

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Khryshchanovich, Study Chair — Educational Institution "Belarusian State Medical University"
Locations (2):
- Belarus (2):
  - Vladimir Khryshchanovich, Minsk, Minsk Oblast
  - Belarusian State Medical University, Minsk

IPD SHARING:
Plan to Share IPD: Yes
To evaluate the clinical efficacy of using graduated compression hosiery for venospecific symptoms, leg edema, and quality of life in pregnant women with varicose veins (VV's).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 05.2022
Access Criteria: To evaluate the clinical efficacy of using graduated compression hosiery for venospecific symptoms, leg edema, and quality of life in pregnant women with varicose veins (VV's).

REFERENCES:
- [Result] Allegra C, Antignani PL, Will K, Allaert F. Acceptance, compliance and effects of compression stockings on venous functional symptoms and quality of life of Italian pregnant women. Int Angiol. 2014 Aug;33(4):357-64. PMID 25056167
- [Result] Gardenghi LA, Dezotti NRA, Dalio MB, Martins WP, Joviliano EE, Piccinato CE. Lower limb venous diameters and haemodynamics during pregnancy and postpartum period in healthy primigravidae. Phlebology. 2017 Dec;32(10):670-678. doi: 10.1177/0268355516671586. Epub 2016 Dec 6. PMID 27928067
- [Result] Smyth RM, Aflaifel N, Bamigboye AA. Interventions for varicose veins and leg oedema in pregnancy. Cochrane Database Syst Rev. 2015 Oct 19;2015(10):CD001066. doi: 10.1002/14651858.CD001066.pub3. PMID 26477632
- [Result] Thaler E, Huch R, Huch A, Zimmermann R. Compression stockings prophylaxis of emergent varicose veins in pregnancy: a prospective randomised controlled study. Swiss Med Wkly. 2001 Dec 1;131(45-46):659-62. doi: 10.4414/smw.2001.09805. PMID 11835115